CLINICAL TRIAL: NCT04766242
Title: The Impact of Spiritual Healing on Moderate Depression in Adults: A Pilot Randomized Controlled Trial (RCT)
Brief Title: The Impact of Spiritual Healing on Moderate Depression in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Tromso (Other)
Collaborators: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 63692
Record Dates: First submitted 2020-11-12; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Moderate Depression
MeSH Terms: interventions — Spiritual Therapies; Touch; Therapeutic Touch

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive 10 healing session of 45-60 minutes as an adjunct to usual care, approximately once a week.The usual care will consist of the treatment plan made by their GP when they were diagnosed with moderate depression.
  Interventions: Other: Spiritual healing; Other: Usual care
- Control group (Other): The control group will receive usual care as prescribed by their GP when they were diagnosed with moderate depression.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Spiritual healing — The spiritual healing will be based on an assessment of the total health situation of the individual patient. Spiritual healing will mainly consist of a treatment where the healers hold their hands for some time at different parts of the patient's body, known as "power points", outside the patients clothing. The consultation might also include possible life-style advice. The treatments will last for 45-60 minutes each time.
  Other Names: Healing touch; Reiki; Hands on healing; Healing by hand; Energy healing
  Arms: Intervention group
Other: Usual care — The care the general practitioner (GP) prescribe when the patients are diagnosed with moderate depression.

SUMMARY:
Depression is a common mental disorder and is together with anxiety the global leading cause of all non-fatal burden of disease. Currently supported treatment for depression is antidepressant medication and different psychotherapeutic interventions. Many patients experience, however, adverse effects of antidepressant medication, while at the same time the access to psychotherapeutic interventions are limited. This is particularly the case for patients suffering from moderate depression. Many patients who suffer from depression turn to complementary and alternative medicine (CAM), and among those therapies often spiritual healing. There is some evidence that consulting a spiritual healer can be beneficial for patients suffer from depression, and that spiritual healing is associated with low risk. The objective of this study is therefor to conduct a pilot RCT (spiritual healing as addition to usual care versus usual care alone) in preparation of a larger trial in adults with moderate depression to examine feasibility and individuals' experience of spiritual healing.

This study is a pilot randomized controlled trial (RCT) with two parallel groups. A total of 28 adult patients with moderate depression according to the M.I.N.I. PLUS DSM-V criteria will be randomized to spiritual healing in addition to usual care intervention (n=14) or usual care alone (n=14). Ten treatment sessions (lasting 45-60 minutes each) of spiritual healing will be administered as an adjunct to usual care and compared to usual care alone. Reduction in depression symptoms will be measured with Beck Depression Inventory (BDI) and Montgomery and Åsberg Depression Rating Scale (MADRS) collected at baseline, week 8 and 16, in addition to BDI measurement collected 6 and 12 months after inclusion in the study. To investigate participants' experience with spiritual healing, a qualitative study will be included using a phenomenological hermeneutical method and semi-structured interviews.

DETAILED DESCRIPTION:
Background Depression is a common mental disorder and is together with anxiety the global leading cause of all non-fatal burden of disease. The core symptoms of depression are lowered mood, discouragement, loss of sense and meaning in life, lack of interest in other people and ordinary duties, and lack of energy and appetite. In addition, often diminished self-esteem, self-reproach and a feeling of guilt. These symptoms may vary in intensity and duration. Nevertheless, around half of people with depression worldwide do not receive treatment. Most mental disorders emerge before the age of 30, and lack of treatment might contribute to disability for many crucial years of an individual's life. In Norway, the 12 months prevalence and lifetime prevalence of depression is 10% and 20% respectably, higher in women than in men. Depression has been identified as a strong predictor for use of complementary and alternative medicine (CAM). A recent Norwegian study demonstrates that only 10.9% of those with moderate depression and/or anxiety visited psychiatric outpatient services while 17.6 % visited a complementary and alternative medicine (CAM) provider. This fact demonstrates that people with depression might be willing to seek help also from less established sources, such as CAM providers. Thus, it is possible that different CAM modalities may serve as a substitute or an alternative when access to psychologist/psychiatric services is limited.

Conventional medicine classifies depression as a mood disorder that manifests itself across a wide range of disease/symptom severity. Depression can be classified as mild, moderate or severe. Symptoms must have been persistent for at least two weeks and not be related to other medical or psychiatric diagnoses, or be due to substances. The World Health Organization ranks the social costs of depression as the 4th highest of all diseases. Furthermore, by 2020 current trends indicate that depression will represent the highest cost to society of any disease. Clearly, prevention, early diagnosis and intervention of depression have huge social significance.

The most commonly prescribed antidepressant drugs, selective serotonin reuptake inhibitors (SSRIs) have recently been shown to have best effect on severe depression, and no effect beyond placebo for mild and moderate depression. At the same time, SSRIs can be associated with serious adverse effects, and are associated with a higher vulnerability to develop a depressive episode later in life. Thus, one of the most common treatment options for depression has been documented to be of little or no help beyond placebo for moderate depression while at the same time possibly inducing serious adverse effects.

The Norwegian minister of health, Bent Høye, has taken the patients' request for an improved treatment situation seriously, and sent a letter to the five regional health authorities in which he wrote: "Many patients in psychological health care do not want to be treated with medication. These patients must be heard and taken seriously. Patients cannot be forced to take medication as long as necessary care and treatment can be provided otherwise".

Cognitive behavioral therapy (CBT) or structured psychological therapy should always be offered patients who do not receive, or do not want pharmaceutical antidepressant treatment. However, the waiting list for such treatments is often long due to the lack of competent professionals (psychologists and psychiatrist), especially in rural communities, but also at the district psychiatric centers are there long waiting lists for such treatments. These centers have to prioritize patients with major depression, meaning that patients with moderate depression have even less access to CBT.

Spiritual healing for depression. Spiritual healing is one of the most frequently used CAM modalities in Norway. It is understood as an energy based therapeutic approach to healing. A spiritual healer uses the hands to balance and harmonies the body and thereby place the client in a position to self-heal. The healing treatment focuses on the whole person (physically, psychologically and emotionally) as well as the environment around the patient. Scientific evidence indicates that users typically praise CAM treatment for offering symptoms relief, reduce side effects of conventional treatment, enhancing their ability to cope physiologically and emotionally, providing an alternative to pharmaceuticals, and offering a close patient-practitioner relationship during treatment.

There is some evidence that spiritual healing can be beneficial for patients suffer from depression and spiritual healing is associated with low risk. In a preliminary study conducted by this current research group, a mean decrease in depression score of 3.1 points (range 0-4) on a 7 point scale was found (n=9). The symptom was rated on a scale from 0-6 where 0 was "as good as it could be "and 6 was "as bad as it could be" (MYMOP scale). Only one patient reported no change in depression symptoms after healing treatment. None of the patients experienced worsening of depression symptoms during the healing treatment while the majority (n=5) had a reduction of 4 points. More research is however needed to confirm these findings and to identify modifications needed in the design of a larger RCT.

Objectives The objectives of this study are to conduct a pilot RCT (spiritual healing as addition to usual care versus usual care alone) in preparation of a larger trial in adults with moderate depression, and further to examine the feasibility of the study design and the participants experience of spiritual healing.

Methods: Pilot RCT with two parallel groups. A total of 28 individuals with moderate depression will be randomized to a spiritual healing intervention as an adjunct to usual care (n=14) or to usual care alone (control) (n=14). In the current study the entire spiritual healing package understood as everything a healer does in a consultation (visiting a healer) will be studied, including the use of hands to balance and harmonies the body and sometimes life style advice. Included in the treatment is the interaction between the patient and the therapist. A positive interaction between the patient and the therapist (alliance) is necessary for the patient to feel free to verbally express painful present and past experiences that may be related to the patient's psychological complaints (e.g., pragmatic research approach).

Informed consent, randomization, control group, allocation concealment: Before the randomization procedures starts, the participants who meet the inclusion criteria and have agreed to participate, read and sign the informed consent after the physician have informed that the participants can withdraw from the study for no reason. The physicians (Arendal and Oslo) will execute the randomisation by drawing sealed opaque envelopes with numbers consecutively from one to 28. Each new patient enrolled in the study will receive the next consecutive envelope, which will be opened after the patient has ended the consultation by the physician, whereas the information about assignment will be known.

A randomisation system with variable block sizes of between two and six will be used, in order to eliminate confounders of a personnel or structural nature, thus balancing group allocation throughout the study period. Within each block, an equal number of patients will be randomly allocated to either an intervention group with spiritual healing and to usual care, or a control group with usual care alone.

Pre-study procedures Patients seeking care for mood related symptoms in Arendal or Oslo will be asked by the physician to participate in the study and screened for possible enrolment. The staff will be oriented about the study procedures and trained before start of the study.

Treatment plan

Spiritual healing The spiritual healing will be based on an assessment of the total health situation of the individual patient. Spiritual healing will mainly consist of a treatment where the healers hold their hands for some time at different parts of the patient's body, known as "power points", outside the patients clothing. The consultation might also include possible life-style advice. This can necessarily lead to slightly different treatment given to each patient. The treatments will, however last for 45-60 minutes each time.

Torunn Anthonsen (Arendal) and Annett Furuseth (Oslo) will perform the healing treatments. The healers are are trained as healers and member of Norwegian healers association (Norges Healerforbund). The healers have worked full time as spiritual healers for more than 5 years. As members of Norwegian healers association, the healers have liability insurance in case of occurrence of harmful events of the treatment.

Usual care Throughout the 16-week intervention period, all participants will be advised to follow the treatment plan given by the physician in Arendal and Oslo. This may include consultation with their physician including life style advices, referral to a psychologist/ psychiatric consultations, anti-depressive medication, and sick leave.

Implementation The study nurse (NAFKAM) will inquire with regard to completeness of prescribed treatment at week 2 and latest at week 16. The patient will also be asked whether he/she has used any other kind of medication, in particular antidepressant medication, visited another health care providers and/or received any other treatment.

Intervention, all patients, stepwise description:

Patients with mood related symptoms who attend the practice of the study physicians in Arendal and Oslo will be asked to participate in a diagnostic interview (conducted by the physician). If the patients meet the inclusion criteria for moderate depression, a treatment plan will be made before randomization to one of the two study groups.

All patients diagnosed with moderate depression according to the M.I.N.I. PLUS DSM-V criteria will be presented to the study and invited to participate until n=28 have accepted the invitation and signed a written consent to participate in the study. 14 participants will be included in Arendal and 14 in in Oslo, (n=7) individuals in intervention group and (n=7) in the control group The physician complete the MADRS baseline questionnaire and the patient complete the BDI baseline questionnaire.

A study nurse (NAFKAM) will then formally include the patient according to the randomisation system with the next envelope in the row.

Included patients will be randomized to spiritual healing plus usual care (intervention group) or usual care alone (control group) Both patients in the intervention group and in the control group are urged to follow the treatment recommendations given by the physician (for example anti-depressant medication or consultations with a psychologist/psychiatrist).

Additional Intervention for the intervention group

Assignment to healing: Name, e-mail address and phone-number of the patients randomized to the intervention group will be delivered (by SMS or email) to the spiritual healer by the research nurse directly after the randomization.

The spiritual healer will contact the patient as soon as possible after the healer have received the name and phone-number.

Patients randomized to the intervention group will get an appointment for healing treatment, and will undergo the first healing session within 2 weeks after inrollment.

The patient will be offered 10 healing sessions. The last follow-up healing treatment session must be completed by the end of week 16 of the study (the day of the first healing session is defined as week 0).

Follow up

At week 8 and 16, the participants and the study physician will complete the BDI and MADR questionnaire. In addition will the participants be asked about adverse effects as part of their form.

Four months after the study inclusion, interviews will be conducted with participants in both groups.

The study nurse (NAFKAM) will contact the participants after 6 and 12 months, and remind the participants to complete the BDI questionnaire (follow-up data). The questionnaire will be forwarded to the participants and will be returned by mail in a pre-payed envelope (figure 1).

Withdrawal and loss to follow-up If a patient chooses to withdraw before week 16, all data collected will be permanently deleted. If the patient is lost to follow-up, data collected up to the day of drop out will be used for analysis.

Statistical analysis Differences in BDI and Madras score between groups as well as adverse effects will be described descriptively only, due to the pilot nature of the study.

Qualitative analysis The qualitative data, will be analyzed using a descriptive qualitative content analysis. Knowledge and understanding of the phenomena under study will be provided through a systematic classification process of coding and identifying themes.

Sample size No sample size calculation is needed for a pilot RCT. A study size of 14 participants in each group is chosen to generate sufficient interviews (saturation on that point is assumed) for the qualitative study. The findings of this pilot study will be used to calculate the sample size in a potential future RCT.

Data handling management All patient data and the index that links trial numbers with individual participants will be kept under lock, and the key will be in the possession of NAFKAM. Trial number alone will identify all data.

Coding and punching Data entry will be undertaken at NAFKAM. Responsible for coding and punching is Agnete Kristoffersen. All data will be read twice to ensure against random bias in the coding and punching process. Trine Stub will be responsible for obtaining and analyze the qualitative data.

Data analysis Data analysis will be done utilizing the IBM statistical package SPSS (http://www.spss.com).

Data and safety monitoring A steering group will be responsible for quality control and meet on a regular basis throughout the study period. The Steering Group will be convened as an emergency in the event of serious adverse effects associated with the trial to decide on appropriate action to prevent recurrence. Regular meetings will concern any reported adverse effects, protocol violation, the recruitment rate, and any practical issues concerning local coordination and the therapists as well as any issues raised by participants.

Ethics and patient safety The patients will be informed about the study through a pamphlet as well as verbally by the study nurse, and, if willing to participate, asked to give a written informed consent. All patients will follow usual care regardless of healing treatment and adverse events will be recorded at each treatment session. No systematic studies have been published on adverse effects of spiritual healing for depression, however, previous research has demonstrated that spiritual healing is associated with low risk. The study will be conducted in accordance with the Helsinki declaration.

The study has been approved by the Regional Committee for Medical and Health Research Ethics (REK 2019/63692). Written informed consent was obtained from all participants.

Study schedule

Provisional milestones

5 of November 2019 Application to the regional ethic committee Winter 2020 Start of inclusion/enrolment/treatment December 2021 Completion of data collection Spring 2022 Data completion and preliminary analysis June 2022 First article sent for publication

Publications The results of the trial are planned to be published in BMC Complementary and Alternative Medicine with the tentative title; "A pilot RCT study with spiritual healing in addition to usual care in the treatment of moderate depression compared to usual care alone".

Organization The research will be based at the National Research Center in Complementary and Alternative Medicine (NAFKAM) in Tromsø, with PI senior researcher Agnete E. Kristoffersen , senior researcher Trine Stub. In addition to study nurse, NAFKAM: Anniken Pettersen and study nurse in Oslo and Arendal, physicians and the spiritual healers: Torunn Anthonsen and Annett Furuseth and psychiatrics and Olav Knudsen-Baas MD, Sørlandet sykehus.

Data and safety monitoring:

A steering group will be responsible for quality control and meet on a regular basis throughout the study period. The Steering Group will be convened as an emergency in the event of serious adverse effects associated with the trial to decide on appropriate action to prevent recurrence. Regular meetings will concern any reported adverse effects, protocol violation, the recruitment rate, and any practical issues concerning local coordination, homeopaths and psychologists, as well as any issues raised by participants.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the criteria for moderate depression
* Have symptoms for two weeks or more
* A minimum of six of the following nine symptoms must have been present:

  1. Depressed mood most of the day
  2. Markedly diminished interest or pleasure in all activities
  3. Significant weight loss or weight gain (more than 5%)
  4. Insomnia or hypersomnia
  5. Psychomotor agitation or retardation
  6. Fatigue
  7. Feelings of worthlessness
  8. Excessive or inappropriate guilt
  9. Diminished ability to concentrate

Minimum one of the six symptoms must be either depressed mood or loss of interest and pleasure.

Exclusion Criteria:

* Symptoms as a direct physiological effects of a substance or a general medical condition
* Substance abuse
* Chronic major or bipolar depression or axis I diagnosis
* Endocrine abnormality; medical disorder or treatment that could cause depression
* Suicidal potential
* Dementia
* Depression due to uncomplicated grief
* History of psychosis or mania
* Heart valve disease
* Poorly controlled hypertension and diabetes mellitus
* Pregnancy
* Inability to complete study forms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the study | through study completion, an average of 2 year".
  • Recruitment speed.
  * The recruitment speed will be recorded in a separate form including the following categories:
    * Dates for first contact with GP
    * Dates for signed consent form
    * Dates for baseline data collection
    * Data for first healing or usual care consultation.
  * Willingness to be randomized will be collected descriptively. The participants will be interviewed about their willingness to be randomized and asked about pros and cons of randomization and input on how to improve the randomization procedure.
  * Study adherence will be collected descriptively. The participants will be interviewed about any obstacles in the study flow and possible improvements.
  * Implementation of healing will be collected descriptively. The participants randomized to healing will be interviewed and asked about the implementation of the healing sessions. The investigators will asked about the participants experiences of the healing treatment (pros and cons).

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) rating scale | Baseline, 8 and 16 weeks
  Change in severity of depression will be measured by Beck Depression Inventory (BDI) rating scale where the participants rate the severity of 21 depression related symptoms raging from 0 to 3 where higher numbers indicate more severe symptoms.
Montgomery and Åsberg Depression Rating Scale (MADRS) | Baseline, 8 and 16 weeks, 6 and 12 months.
  Change in severity of the participants depression measured by Montgomery and Åsberg Depression Rating Scale (MADRS) where the physician rate 10 depression related symptoms on a scale from 0 to 6 where higher numbers indicate more severe symptoms
Semi-structured interviews | 16 weeks after first participant enrollment until 16 weeks after the last participant has been enroled in the study.
  Nested within the RCT the investigators will perform interviews with the participants to investigate participants' experience of spiritual healing and the study design using a phenomenological Hermeneutical method and semi-structured interviews. In this qualitative study the participants will be encouraged to tell their own study as participants in the present RCT. They will be questioned about their expectations to the study and whether these expectations were meet. The investigators will also asked them what worked (e.g. requirement, randomization procedures, blinding and how they experienced the healing and usual care sessions) and what did not work. In this qualitative study the outcome will be collected as text data and no scales will be used. The data will be analyzed descriptively (content analysis).

OTHER OUTCOMES:
Adverse effects of the treatment | All through the study
  During the intervention period, the health care providers will ask specifically about, and record any adverse effect of the treatment that may have occurred since last consultation and adverse effect forms will be completed after 8 and 16 weeks. The Relis adverse effect scale will be used to measure adverse effects (35). For reporting of adverse effects of healing treatment, a modified adverse effect form will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Uit The Arctic University of Norway, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whiteford HA, Degenhardt L, Rehm J, Baxter AJ, Ferrari AJ, Erskine HE, Charlson FJ, Norman RE, Flaxman AD, Johns N, Burstein R, Murray CJ, Vos T. Global burden of disease attributable to mental and substance use disorders: findings from the Global Burden of Disease Study 2010. Lancet. 2013 Nov 9;382(9904):1575-86. doi: 10.1016/S0140-6736(13)61611-6. Epub 2013 Aug 29. PMID 23993280
- [Background] Wang PS, Aguilar-Gaxiola S, Alonso J, Angermeyer MC, Borges G, Bromet EJ, Bruffaerts R, de Girolamo G, de Graaf R, Gureje O, Haro JM, Karam EG, Kessler RC, Kovess V, Lane MC, Lee S, Levinson D, Ono Y, Petukhova M, Posada-Villa J, Seedat S, Wells JE. Use of mental health services for anxiety, mood, and substance disorders in 17 countries in the WHO world mental health surveys. Lancet. 2007 Sep 8;370(9590):841-50. doi: 10.1016/S0140-6736(07)61414-7. PMID 17826169
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Eisenberg D, Golberstein E, Gollust SE. Help-seeking and access to mental health care in a university student population. Med Care. 2007 Jul;45(7):594-601. doi: 10.1097/MLR.0b013e31803bb4c1. PMID 17571007
- [Background] Druss BG, Rosenheck RA. Use of practitioner-based complementary therapies by persons reporting mental conditions in the United States. Arch Gen Psychiatry. 2000 Jul;57(7):708-14. doi: 10.1001/archpsyc.57.7.708. PMID 10891042
- [Background] Kessler RC, Soukup J, Davis RB, Foster DF, Wilkey SA, Van Rompay MI, Eisenberg DM. The use of complementary and alternative therapies to treat anxiety and depression in the United States. Am J Psychiatry. 2001 Feb;158(2):289-94. doi: 10.1176/appi.ajp.158.2.289. PMID 11156813
- [Background] Spinks J, Hollingsworth B. Policy implications of complementary and alternative medicine use in Australia: data from the National Health Survey. J Altern Complement Med. 2012 Apr;18(4):371-8. doi: 10.1089/acm.2010.0817. PMID 22515796
- [Background] Hansen AH, Kristoffersen AE. The use of CAM providers and psychiatric outpatient services in people with anxiety/depression: a cross-sectional survey. BMC Complement Altern Med. 2016 Nov 11;16(1):461. doi: 10.1186/s12906-016-1446-9. PMID 27835971
- [Background] Bazargan M, Ani CO, Hindman DW, Bazargan-Hejazi S, Baker RS, Bell D, Rodriquez M. Correlates of complementary and alternative medicine utilization in depressed, underserved african american and Hispanic patients in primary care settings. J Altern Complement Med. 2008 Jun;14(5):537-44. doi: 10.1089/acm.2007.0821. PMID 18537468
- [Background] Jorm AF, Griffiths KM, Christensen H, Parslow RA, Rogers B. Actions taken to cope with depression at different levels of severity: a community survey. Psychol Med. 2004 Feb;34(2):293-9. doi: 10.1017/s003329170300895x. PMID 14982135
- [Background] MacPherson H, Thorpe L, Thomas K, Geddes D. Acupuncture for depression: first steps toward a clinical evaluation. J Altern Complement Med. 2004 Dec;10(6):1083-91. doi: 10.1089/acm.2004.10.1083. PMID 15674005
- [Background] Kirsch I, Deacon BJ, Huedo-Medina TB, Scoboria A, Moore TJ, Johnson BT. Initial severity and antidepressant benefits: a meta-analysis of data submitted to the Food and Drug Administration. PLoS Med. 2008 Feb;5(2):e45. doi: 10.1371/journal.pmed.0050045. PMID 18303940
- [Background] Arroll B, Elley CR, Fishman T, Goodyear-Smith FA, Kenealy T, Blashki G, Kerse N, Macgillivray S. Antidepressants versus placebo for depression in primary care. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD007954. doi: 10.1002/14651858.CD007954. PMID 19588448
- [Background] Van Aken R, Taylor B. Emerging from depression: the experiential process of Healing Touch explored through grounded theory and case study. Complement Ther Clin Pract. 2010 Aug;16(3):132-137. doi: 10.1016/j.ctcp.2009.11.001. Epub 2009 Dec 5. PMID 20621272
- [Background] Shore AG. Long-term effects of energetic healing on symptoms of psychological depression and self-perceived stress. Altern Ther Health Med. 2004 May-Jun;10(3):42-8. PMID 15154152
- [Background] Richeson NE, Spross JA, Lutz K, Peng C. Effects of Reiki on anxiety, depression, pain, and physiological factors in community-dwelling older adults. Res Gerontol Nurs. 2010 Jul;3(3):187-99. doi: 10.3928/19404921-20100601-01. Epub 2010 Jun 30. PMID 20635803
- [Background] Joyce J, Herbison GP. Reiki for depression and anxiety. Cochrane Database Syst Rev. 2015 Apr 3;2015(4):CD006833. doi: 10.1002/14651858.CD006833.pub2. PMID 25835541
- [Background] Kristoffersen AE, Stub T, Knudsen-Baas O, Udal AH, Musial F. Self-Reported Effects of Energy Healing: A Prospective Observational Study With Pre-Post Design. Explore (NY). 2019 Mar-Apr;15(2):115-125. doi: 10.1016/j.explore.2018.06.009. Epub 2018 Aug 22. PMID 30262161
- [Background] Paterson C, Britten N. In pursuit of patient-centred outcomes: a qualitative evaluation of the 'Measure Yourself Medical Outcome Profile'. J Health Serv Res Policy. 2000 Jan;5(1):27-36. doi: 10.1177/135581960000500108. PMID 10787584
- [Background] Thompson TD, Weiss M. Homeopathy--what are the active ingredients? An exploratory study using the UK Medical Research Council's framework for the evaluation of complex interventions. BMC Complement Altern Med. 2006 Nov 13;6:37. doi: 10.1186/1472-6882-6-37. PMID 17101037
- [Background] Pennebaker JW, Barger SD, Tiebout J. Disclosure of traumas and health among Holocaust survivors. Psychosom Med. 1989 Sep-Oct;51(5):577-89. doi: 10.1097/00006842-198909000-00009. PMID 2798704
- [Background] Steer RA, Cavalieri TA, Leonard DM, Beck AT. Use of the Beck Depression Inventory for Primary Care to screen for major depression disorders. Gen Hosp Psychiatry. 1999 Mar-Apr;21(2):106-11. doi: 10.1016/s0163-8343(98)00070-x. PMID 10228890
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Derived] Stub T, Irgens AC, Hansen AH, Knudsen-Baas O, Gaskjenn C, Kristoffersen AE. Impact of spiritual healing on moderate depression in adults: a study protocol of a pilot randomised controlled trial (RCT). BMJ Open. 2022 Sep 15;12(9):e062683. doi: 10.1136/bmjopen-2022-062683. PMID 36109024
- See also: Medikamentfri behandling for psykiske syke i alle helseregioner — https://www.regjeringen.no/no/aktuelt/medikamentfri-behandling-for-psykisk-syke-i-alle-helseregioner/id2464240/.
- See also: Depression — https://helsedirektoratet.no/folkehelse/psykisk-helse-og-rus/angst-og-depresjon/depresjon
- See also: The use of complementary and alternative medicine (CAM) in Norway, 2018 — https://nafkam.no/sites/default/files/2019-06/NAFKAM-2018%20report%20EN%20%28002%29_0.pdf
- See also: Diagnostic and Statistical Manual of Mental Disorders (DSM-5) American Psychiatric Association — https://psychiatry.org/psychiatrists/practice/dsm
- See also: Notice of suspected adverse reaction when using medicines (including herbal medicines) — http://www.legemiddelverket.no